CLINICAL TRIAL: NCT00650923
Title: Phase I Trial of Aflibercept (VEGF Trap) With Radiation Therapy and Concomitant and Adjuvant Temozolomide in Patients With Malignant Glioma
Brief Title: Aflibercept, Radiation Therapy, and Temozolomide in Treating Patients With Newly Diagnosed or Recurrent Glioblastoma Multiforme, Gliosarcoma, or Other Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00678; NCI-2009-00678 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000590174; NABTC-07-01; NABTC07-01 (Other: Adult Brain Tumor Consortium); NABTC-07-01 (Other: CTEP); U01CA137443 (NIH)
Record Dates: First submitted 2008-04-01; First posted 2008-04-02 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-04

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — aflibercept; Radiotherapy; Radiation; Temozolomide

ARMS (1):
- Arm 1 (Experimental): See Detailed Description
  Interventions: Drug: ziv-aflibercept; Procedure: radiation therapy; Drug: temozolomide; Procedure: pharmacological study; Procedure: laboratory biomarker analysis

INTERVENTIONS:
Drug: ziv-aflibercept — Given IV
  Other Names: aflibercept; vascular endothelial growth factor trap; VEGF Trap; Zaltrap
Procedure: radiation therapy — Undergo RT
  Other Names: irradiation; radiotherapy; therapy, radiation
Drug: temozolomide — Given PO
  Other Names: SCH 52365; Temodal; Temodar; TMZ
Procedure: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Procedure: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of aflibercept when given together with radiation therapy and temozolomide in treating patients with newly diagnosed or recurrent glioblastoma multiforme, gliosarcoma, or other malignant glioma. Aflibercept may stop the growth of tumor cells by blocking blood flow to the tumor. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving aflibercept together with radiation therapy and temozolomide may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the maximum tolerated dose (MTD) of aflibercept (VEGF Trap) with radiotherapy (RT) and concurrent temozolomide (TMZ) when administered in patients with newly-diagnosed glioblastoma (GBM) or gliosarcoma.

II. To define the MTD of aflibercept with adjuvant TMZ administered at 150mg/m2once daily for 5 days every 28 days in patients with stable or recurrent malignant glioma (MG) after RT.

III. To define the MTD of aflibercept with adjuvant TMZ administered at 100 mg/m2 once daily for 21 days every 28 days in patients with stable or recurrent MG after RT.

IV. To characterize the safety profile of aflibercept in combination with RT and concomitant TMZ in patients with newly-diagnosed GBM.

V. To characterize the safety profile of aflibercept in combination with adjuvant TMZ in patients with stable or recurrent MG after RT.

SECONDARY OBJECTIVE:

I. To characterize the pharmacokinetic profiles of free and bound aflibercept and TMZ in these patients

OUTLINE: This is a multicenter, dose-escalation study of aflibercept. Patients are assigned to 1 of 3 treatment groups according to prior treatment and diagnosis.

Group 1 (newly diagnosed glioblastoma multiforme or gliosarcoma): Patients undergo involved field partial brain radiotherapy (RT) once daily, 5 days a week (total of 30 fractions) and receive concurrent oral temozolomide (TMZ) once daily for 6 weeks. Beginning 2 weeks after the initiation of RT patients also receive aflibercept IV over 1 hour on days 1 and 15 and continue until the end of RT. Beginning 4 weeks after completion of radiotherapy, patients receive adjuvant oral TMZ once daily on days 1-5. Treatment with adjuvant TMZ repeats every 28 days for up to 12 courses.

Group 2 (stable or recurrent malignant glioma): Patients undergo radiotherapy as in group 1. Patients receive oral TMZ on days 1-5. Treatment repeats every 28 days for up to 12* courses. Patients also receive aflibercept IV over 1 hour on days 1 and 15 beginning on the first day of TMZ treatment.

[Note: *The 12 course maximum includes adjuvant TMZ courses administered prior to enrollment.]

Group 3 (stable or recurrent malignant glioma): Patients undergo radiotherapy as in group 1. Patients receive oral TMZ on days 1-5. Treatment repeats every 21 days for up to 12* courses. Patients also receive aflibercept IV over 1 hour on days 1 and 15 beginning on the first day of TMZ treatment.

[Note: *The 12 course maximum includes adjuvant TMZ courses administered prior to enrollment.]

In all groups, treatment continues in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for analysis of pharmacokinetics by ELISA. Tumor biomarkers and plasma angiogenic peptides are analyzed for correlation with response, and tumor MGMT promoter methylation status is determined using methylation-specific PCR.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
Criteria:

* Creatinine < = 1.5 mg/dL or creatinine clearance = > 60 mL/min
* At least 28 days since prior major surgery or open biopsy
* INR < = 1.5
* Not pregnant or nursing
* Negative pregnancy test
* Karnofsky performance status 60-100%
* SGOT and SGPT < 2 times upper limit of normal (ULN)
* Bilirubin < 2 times ULN
* Life expectancy = > 12 weeks
* WBC = > 3,000/μL
* ANC= > 1,500/mm³
* Platelet count = > 100,000/mm³
* Hemoglobin = > 10 g/dL (transfusion allowed)
* At least 21 days since prior radiotherapy (groups 2 and 3)
* No prior Gliadel® wafers
* No concurrent major surgery
* Fertile patients must use effective contraception prior to, during, and for at least 6 months after completion of study treatment
* At least 28 days since prior significant traumatic injury No evidence of bleeding diathesis or coagulopathy
* No serious or nonhealing wound, ulcer, or bone fracture
* No history of other cancer (except nonmelanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years
* No history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess gastrointestinal bleeding or diverticulitis within the past 6 months
* No prior cranial radiotherapy (group 1 only)
* No prior aflibercept
* No prior treatment for brain tumors, except concurrent radiotherapy and temozolomide or 2 or fewer 28-day courses of adjuvant temozolomide (groups 2 and 3)
* No prior or concurrent cytotoxic drug therapy, non-cytotoxic drug therapy, or experimental drug therapy for brain tumors (group 1 only)
* No concurrent major surgery
* No known hypersensitivity to CHO cell products or other recombinant human antibodies
* No history of hypersensitivity to a recombinant protein whereby reaction occurs during or immediately after infusion
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to other study agents
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness or social situation that would limit compliance with study requirements
* No clinically significant cardiovascular disease within the past 6 months, including any of the following:

History of ischemic or hemorrhagic stroke

* Myocardial infarction, coronary artery bypass graft, or unstable angina
* New York Heart Association class III-IV congestive heart failure, serious cardiac arrhythmia requiring medication, or unstable angina pectoris
* Clinically significant peripheral vascular disease
* Pulmonary embolism, deep vein thrombosis, or other thromboembolic event
* No disease that will obscure toxicity or dangerously alter drug metabolism
* Recovered from all prior therapy
* More than 28 days since prior and no concurrent investigational agents
* More than 7 days since prior core biopsy
* At least 23 days since prior temozolomide (groups 2 and 3)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent full-dose anticoagulants (e.g., warfarin or low molecular-weight heparin)
* Prophylactic doses allowed
* No concurrent routine prophylactic use of filgrastim (G-CSF)
* No other concurrent anticancer therapy (including chemotherapy, radiotherapy, hormonal treatment, or immunotherapy)
* Concurrent enzyme-inducing antiepileptic drugs (EIAED) or non-EIAED allowed
* Urine protein:creatinine ratio < = 1 or 24-hour urine protein < = 500 mg
* No significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-07; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of aflibercept defined as the dose at which fewer than one-third of patients experience DLT based on the CTC severity grading | 28 days

SECONDARY OUTCOMES:
Efficacy in terms of antitumor activity based on clinical, radiographic, and biologic assessments | Up to 3 months
  Descriptive analysis will be provided.
Plasma aflibercept (VEGF Trap) concentrations and PK parameters such as Cmax, Tmax, area under the plasma concentration-time curve (AUCo-t and AUC), clearance (CL), apparent volume of distribution at steady state (Vdss), and terminal half-life (t1/2) | Baseline and days 15, 16, 22, 29, 57, 85 of course 1 for patients in Arm I; baseline and days 2, 8, 15, 43, 71 of course 1 for patients in Arms 2 and 3
  Will be determined using non-compartmental methods. Dose proportionality in PK parameters will be determined by performing a one-way analysis of variance (ANOVA) on dose-normalized parameters. In addition, summary tables depicting individual patient concentrations and individual and mean PK parameters will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wen, Principal Investigator — National Cancer Institute (NCI)
Locations (9):
- United States (9):
  - University of California at Los Angeles (UCLA ), Los Angeles, California
  - UCSF-Mount Zion, San Francisco, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Adult Brain Tumor Consortium, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas